CLINICAL TRIAL: NCT04587713
Title: A Phase 1, Two-Part, Open-Label Study to Assess the Relative Bioavailability of Two TD-1473 Tablet Formulations Under Fasted and Fed Conditions in Healthy Subjects and the Pharmacokinetics of TD-1473 in Healthy Chinese Subjects
Brief Title: Single Dose Bioavailability and Ethnobridging PK Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0184
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Intestinal Disorder; Bowel Diseases, Inflammatory
Keywords: Healthy Caucasian Subjects; Healthy Chinese Subjects; Ethnobridging
MeSH Terms: conditions — Intestinal Diseases; Inflammatory Bowel Diseases | interventions — izencitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A, Sequence 1 (Experimental): Part A, Sequence 1 = Treatment (Tx) C, Tx A, Tx C, Tx A
  Single oral dose of treatment on Day 1 of each period in a 4-way crossover design with a ≥10-day washout between treatments
  Interventions: Drug: TD-1473 [Tablet A]; Drug: TD-1473 [Tablet B]
- Part A, Sequence 2 (Experimental): Part A, Sequence 2: Tx D, Tx B, Tx D, Tx B
  Single oral dose of treatment on Day 1 of each period in a 4-way crossover design with a ≥10-day washout period between treatments
  Interventions: Drug: TD-1473 [Tablet A]; Drug: TD-1473 [Tablet B]
- Part A, Sequence 3 (Experimental): Part A, Sequence 3: Tx C, Tx A, Tx D, Tx B
  Single oral dose of treatment on Day 1 of each period in a 4-way crossover design with a ≥10-day washout period between treatments
  Interventions: Drug: TD-1473 [Tablet A]; Drug: TD-1473 [Tablet B]
- Part A, Sequence 4 (Experimental): Part A, Sequence 4: Tx D, Tx B, Tx C, Tx A
  Single oral dose of treatment on Day 1 of each period in a 4-way crossover design with a ≥10-day washout period between treatments
  Interventions: Drug: TD-1473 [Tablet A]; Drug: TD-1473 [Tablet B]
- Part A, Sequence 5 (Experimental): Part A, Sequence 5: Tx A, Tx C, Tx A, Tx C
  Single oral dose of treatment on Day 1 of each period in a 4-way crossover design with a ≥10-day washout period between treatments
  Interventions: Drug: TD-1473 [Tablet A]; Drug: TD-1473 [Tablet B]
- Part A, Sequence 6 (Experimental): Part A, Sequence 6: Tx B, Tx D, Tx B, Tx D
  Single oral dose of treatment on Day 1 of each period in a 4-way crossover design with a ≥10-day washout period between treatments
  Interventions: Drug: TD-1473 [Tablet A]; Drug: TD-1473 [Tablet B]
- Part A, Sequence 7 (Experimental): Part A, Sequence 7: Tx A, Tx C, Tx B, Tx D
  Single oral dose of treatment on Day 1 of each period in a 4-way crossover design with a ≥10-day washout period between treatments
  Interventions: Drug: TD-1473 [Tablet A]; Drug: TD-1473 [Tablet B]
- Part A, Sequence 8 (Experimental): Part A, Sequence 8: Tx B, Tx D, Tx A, Tx C
  Single oral dose of treatment on Day 1 of each period in a 4-way crossover design with a ≥10-day washout period between treatments
  Interventions: Drug: TD-1473 [Tablet A]; Drug: TD-1473 [Tablet B]
- Part B,Treatment A (Experimental): Single oral dose of Treatment A on Day 1
  Interventions: Drug: TD-1473 [Tablet A]

INTERVENTIONS:
Drug: TD-1473 [Tablet A] — TD-1473 [Tablet A] (1 Tablet = Dose A) proposed commercial tablet formulation
Drug: TD-1473 [Tablet B] — TD-1473 [Tablet B] (2 Tablets = Dose A) current clinical tablet formulation
  Arms: Part A, Sequence 1; Part A, Sequence 2; Part A, Sequence 3; Part A, Sequence 4; Part A, Sequence 5; Part A, Sequence 6; Part A, Sequence 7; Part A, Sequence 8

SUMMARY:
This is a Phase 1, 2-part, open-label study. Part A will be a formulation bridging and food effect study in healthy adult subjects. Part B will be an assessment of pharmacokinetics (PK) in healthy adult Chinese subjects.

DETAILED DESCRIPTION:
In study Part A, healthy adult subjects will receive the following treatments in a cross-over design with a ≥10-day washout period between doses:

* Treatment A: Single dose of [Tablet A] TD-1473 proposed commercial tablet formulation on Day 1 in a fasted state;
* Treatment B: Single dose of [Tablet A] TD-1473 proposed commercial tablet formulation on Day 1 in a fed state;
* Treatment C: Single dose of [Tablet B] TD-1473 current clinical tablet formulation on Day 1 in a fasted state;
* Treatment D: Single dose of [Tablet B] TD-1473 current clinical tablet formulation on Day 1 in a fed state.

In study Part B, healthy adult Chinese subjects will receive Treatment A: Single dose of [Tablet A] TD-1473 proposed commercial tablet formulation on Day 1 in a fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a non-smoking male or female adult
* Subject (females) must be of non-childbearing potential or if of childbearing potential, subject must not be pregnant or breastfeeding, and must agree to use highly effective birth control and must not donate ova through 30 days after last dose of study drug.
* Subject (males) must agree to use contraception to prevent pregnancy/partner exposure and must not donate sperm through 30 days after last dose of study drug.
* Subject has a body mass index (BMI) 19 to 30 kg/m^2, inclusive and weighs at least 50 kg
* Subject is healthy as determined by the Principal Investigator or designee based on medical history and physical examinations performed at Screening and Day -1 of Period 1
* Subject must be willing and able to comply with the study diet, willing to abstain from strenuous physical activity which could cause muscle aches or injury, including contact sports for a period of 48 hours prior to study and through follow-up visit.
* Subject must be willing and able to give and understand written informed consent, communicate well with the PI, and comply with the study procedures, requirements and restrictions
* Part B: subject was born in China, with 2 Chinese biological parents and 4 Chinese grandparents as confirmed by interview, has lived no longer than 10 years outside of China, and has had no significant change in lifestyle, including diet, since leaving China

Exclusion Criteria:

* Subject is planning to conceive a child during the study or within 1 month after the last dose of TD 1473
* Subject has evidence or history of clinically significant allergic disease, hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease
* Subject has history of venous thrombosis
* Subject has any clinically significant abnormalities in the results of laboratory evaluations, or liver function tests exceeding the upper limit of normal in the screening or pre-dose period
* Subject has creatinine clearance as calculated by Cockcroft-Gault formula <90mL/min at screening or pre-dose period.
* Subject has any medical condition possibly affecting drug absorption
* Subject has history of lymphoma, leukemia, or other types of malignancy
* Subject previously participated in a study for TD 1473 and/or subject has previously taken tofacitinib or other JAK inhibitors.
* Subject participated in another clinical trial of an investigational drug (or medical device) within 30 days
* Subject is unwilling to abstain from ingestion of caffeine or xanthine-containing products
* Subject is unwilling to abstain from alcohol beginning 24 hours prior to study start
* Subject has history of alcoholism or drug abuse
* Female subject who is pregnant and/or lactating
* Subject has positive results at Screening for human immunodeficiency virus (HIV), hepatitis A virus (HAV) antibodies, hepatitis B virus antigen (HBsAg), hepatitis B core antibodies (HBcAb), or hepatitis C virus (HCV) antibody
* Subject has confirmed or suspected severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection (COVID-19)
* Subject consumed grapefruit/Seville orange and/or grapefruit juice within 14 days prior to study
* Subject consumed cruciferous vegetables (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard greens) or charbroiled meats beginning 7 days prior to study start and is unwilling to abstain from consuming such vegetables during the study
* Subject uses or has used nicotine-containing products within 6 months prior to study start
* Subject has acute illness (GI illness, infection (e.g., influenza) or know inflammatory process) at screening or pre-dose period.
* Subject has poor venous access that limits phlebotomy
* Subject donated blood or had significant blood loss within 56 days prior to study start
* Subject donated plasma within 7 days prior to study start
* Subject has abnormal screening ECG based on certain parameters or designated by the PI or designee to be clinically significant.
* Subject has personal or known family history of congenital long QT syndrome or known family history of sudden death
* Subject has history of hypersensitivity to drugs with a clinically significant reaction or any clinically significant hypersensitivities
* Subject has known hypersensitivity to contents of the study drug including excipients, or drugs from a similar chemical class as TD-1473
* Subject has history of severe allergic reaction or severe hypersensitivity or idiosyncratic reaction to any food, medication, insect or bee sting, or previous status asthmaticus (e.g., acute severe asthma attacks)
* Subject has history of latent or active tuberculosis
* Subject received a live viral vaccine within 8 weeks of study start
* Subject, who, for any reason, is deemed by the Principal Investigator, designee, or Sponsor to be inappropriate for this study or have any condition which would confound or interfere with the evaluation of the safety, tolerability, and PK of the investigational drug or prevent compliance with the study protocol

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-27 (Actual)

PRIMARY OUTCOMES:
AUC0-t | Predose and at prespecified time points up to 5 days after dosing on Day 1 of each period
  Area under the concentration-time curve, from time 0 to the last observed non-zero concentration (AUC0-t) of TD-1473 in Plasma
AUC0-inf | Predose and at prespecified time points up to 5 days after dosing on Day 1 of each period
  Area under the concentration-time curve, from time 0 extrapolated to infinity (AUC0-inf) of TD-1473 in Plasma
Cmax | Predose and at prespecified time points up to 5 days after dosing on Day 1 of each period
  Maximum observed concentration (Cmax) of TD-1473 in Plasma

SECONDARY OUTCOMES:
Adverse events | Day 1 through Day 7 of each period
  Number and severity of treatment emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Theravance Biopharma
Locations (2):
- United States (2):
  - Theravance Biopharma Investigational Site, Cypress, California
  - Theravance Biopharma Investigational Site, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.